CLINICAL TRIAL: NCT02197325
Title: Pressure Controlled Intermittent Coronary Sinus Occlusion (PiCSO) as an Adjunct to PCI in Acute Coronary Syndrome
Brief Title: PiCSO in ACS Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miracor Medical SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP2014-03
Record Dates: First submitted 2014-07-16; First posted 2014-07-22 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Acute Coronary Syndrome
Keywords: NSTEMI and STEMI
MeSH Terms: conditions — Acute Coronary Syndrome; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PICSO (Active Comparator): Participants enrolled in the PICSO treatment Group will be treated with PICSO concomitant to pPCI in patients with anterior non ST-segment Elevation Myocardial Infarction or following pPCI in ST-segment Elevation Myocardial Infarction
  Interventions: Device: PICSO
- Parallel control (No Intervention): Participants enrolled in will receive treatment based on the standard guidelines for treatment of a myocardial infarction.

INTERVENTIONS:
Device: PICSO — Pressure controlled Intermittent Coronary Pressure Occlusion
  Other Names: PICSO Impulse System
  Arms: PICSO

SUMMARY:
The purpose of this research study is to find out whether PICSO (Pressure Controlled Coronary Sinus Occlusion), given concomitant to (NSTEMI) or following (STEMI) primary PCI and stenting, can improve final infarct size and myocardial function.

ACS patients, NSTEMI and STEMI, with a culprit lesion in the LAD will be treated according to standard treatment, PCI followed by stent placement, with or without PICSO therapy. In NSTEMI patients, PICSO therapy will be given during PCI and stenting for a minimum of 30 minutes or the duration of the PCI and stent procedure. In STEMI patients PICSO therapy will be given after successful primary percutaneous coronary intervention of a left anterior descending coronary artery culprit lesion. PICSO therapy is initiated prior to stent deployment and continued during stenting. The functional efficacy measures, related to the PICSO duration and coronary sinus pressures, will be stored on the PICSO Impulse console and analysed offline. The clinical efficacy measures, cardiac enzyme release during 24 hour following PCI, cardiac function, infarct size and level of microvascular obstruction will be assessed by cMRI. Patients will be followed for a maximum of 4 months after the primary PCI procedure

DETAILED DESCRIPTION:
The study is designed to evaluate the effect of PICSO treatment concomitant to or following primary PCI in patients with anterior non ST-segment Elevation Myocardial Infarction or ST-segment Elevation Myocardial Infarction, in patients with a culprit lesion in the LAD on Infarct Size and myocardial function. There will be 2 phases in this study.

1. Phase 1: only NSTEMI patients will be recruited.
2. Phase 2: only STEMI patients will be recruited.

Phase 1 During Phase 1 of the study only NSTEMI patients will be recruited. After having given informed consent the patient will be scheduled for pPCI and stent placement. On the day of the procedure the PICSO catheter will be placed as described below (refer to PICSO Impulse catheter placement). After the PICSO therapy is started the standard pPCI and stent placement is performed. PICSO is continued at a minimum of 30 minutes or as long as the standard pPCI and stent placement takes.

Phase 2 During Phase 2 of the study only STEMI patients will be recruited. Immediately after successful restoration of the blood flow the PICSO Impulse catheter is introduced and placed as described below (Refer to PICSO Impulse catheter placement).

After correct positioning of the PICSO Impulse catheter, the 0,032" guide wire is removed. PICSO therapy is initiated and continued until a PICSO Quantity of 1000 mmHg is reached or a maximum of 60 minutes active treatment whatever comes first. With PICSO in treatment mode, the stent is deployed.

The clinical outcome data collected will be based on the site standards of care for NSTEMI and acute STEMI. Examinations include but are not limited to physical assessments, cardiac markers, ECG, laboratory results, x-rays, angiograms, cMRI and echocardiography.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with first time symptoms of acute coronary syndrome (NSTEMI and STEMI)
2. Culprit lesion in the LAD.
3. Age range 25 - 75 years

Exclusion Criteria:

1. Complicated PCI of an LAD culprit lesion (defined as angioplasty followed by stent placement or direct stenting with the occurrence of an adverse event(s) that would preclude further interventional procedures during the index procedure, such as major bleeding, perforation, hypotension, pulmonary edema or instability that in the judgment of the investigator precludes use of the PICSO Impulse System).
2. Previous coronary artery bypass graft surgery
3. History of stroke, TIA or reversible ischemic neurological disease within last 6 months
4. Hospitalization with a primary diagnosis of acute myocardial infarction (AMI) previously or has evidence of previous Q-wave infarct
5. Known contra-indication for magnetic resonance imaging (Metallic implant precluding MRI, claustrophobia, obesity precluding MRI, etc.)
6. Active or treated malignancies in the last 12 months
7. Pregnant Women
8. Non-cardiac comorbidities and life expectancy < 1 year
9. Use of warfarin

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2015-01; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in Infarct Size assessed by cardiac MRI | baseline and 4 months
  Efficacy of PICSO treatment as assessed by means of infarct size reduction assessment, 4-months vs. 1 week post-primary PCI in comparison with a matched non-PICSO parallel control group

SECONDARY OUTCOMES:
Enzymatic Infarct Size | 12 hours post PCI
  Peak Troponin level 12 hours after pPCI, in comparison with a matched non-PICSO parallel control group
Level of Microvascular Obstruction assessed by cardia MRI | 2-5 days post PCI
  Microvascular Obstruction assessed by cardiac MRI on 2-5 days post pPCI
Absolute Infarct size assessment by cardiac MRI | baseline and 4 months
  Infarct size assessment by cardiac MRI (presented as % of Area at Risk, AAR, and % of LV) at 2-5 days and 120 ± 14 days post-primary PCI in comparison with a matched non-PICSO parallel control group.
MACE | baseline to 4 months
  Occurrence of major adverse cardiac events (MACE) during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Azfar Zaman, Prof. Dr., Principal Investigator — Freeman Hospital, Newcastle
Locations (4):
- United Kingdom (4):
  - Liverpool Heart and Chest Hospital, Liverpool
  - St Bartholomew's Hospital, London
  - Freeman Hospital, Newcastle
  - Northern General Hospital, Sheffield